CLINICAL TRIAL: NCT02657525
Title: Acute Exacerbation of Chronic Obstructive Pulmonary Disease Inpatient Registry Study
Acronym: AECOPD-IRS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Peking University (Other); China Soong Ching Ling Foundation (Other)
Responsible Party: Principal Investigator, Chen Wang, Prof.Dr., China-Japan Friendship Hospital
Other Study IDs: 2015-88
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the demographic characteristics, clinical features, diagnoses and treatments of AECOPD hospitalized patients in China, and disease prognosis and its economic burden.

ELIGIBILITY:
Inclusion Criteria:

≥18 years of age; hospitalized patients with main diagnosis as AECOPD.

Exclusion Criteria:

Patients diagnosed as active pulmonary tuberculosis, or acute left heart failure; Patients participating in clinical trials or intervention studies of drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AECOPD-IRS plans to enroll 7600 hospitalized patients (≥ 18 years old with main diagnosis as AECOPD). Sample size estimation is based on estimated mortality of AECOPD hospitalized patients (~5%). Study patients will be recruited from 40-60 hospitals across China,each hospital will recruit 152-190 patients. Hospital selection follows a multi-stage sampling strategy.
Sampling Method: Probability Sample
Enrollment: 7600 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 12 months
  All-cause and cause-specific mortality will be described.
Readmission | 12 months
  Readmission rate caused by AECOPD within 1 month after discharged from hospital.

SECONDARY OUTCOMES:
All-cause and cause-specific mortality | 3 years
  All-cause and cause-specific mortality will be described at different time points (1, 2, 3 years)
Recurrence of acute exacerbation of COPD | 3 years
  Frequency of AECOPD recurrence will be described during follow-ups, the date of first recurrence after discharge will be analysed.
Lung function and quality of life assessment | 3 years
  Lung function will be measured regularly, quality of life will be assessed by questionnaires
Healthcare costs | 12 months
  Direct costs of hospital stay will be recorded.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Niu Y, Niu H, Meng X, Zhu Y, Ren X, He R, Wu H, Yu T, Zhang Y, Kan H, Chen R, Yang T, Wang C. Associations Between Air Pollution and the Onset of Acute Exacerbations of COPD: A Time-Stratified Case-Crossover Study in China. Chest. 2024 Nov;166(5):998-1009. doi: 10.1016/j.chest.2024.05.030. Epub 2024 Jun 19. PMID 38906462
- [Derived] He R, Wang Y, Ren X, Huang K, Lei J, Niu H, Li W, Dong F, Li B, Yang T, Wang C. Associations of medication regimen complexity with medication adherence and clinical outcomes in patients with chronic obstructive pulmonary disease: a prospective study. Ther Adv Respir Dis. 2023 Jan-Dec;17:17534666231206249. doi: 10.1177/17534666231206249. PMID 37855117